CLINICAL TRIAL: NCT01301586
Title: A RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO ASSESS THE SAFETY AND EFFICACY OF A NOVEL ORAL ACNE TREATMENT FOR THE TREATMENT OF ACNE VULGARIS
Brief Title: A Novel Combination Oral Agent to Treat Acne Vulgaris
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nexgen Dermatologics, Inc. (Industry)
Responsible Party: H. Gary Berlin, Nexgen Dermatologics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11022006
Record Dates: First submitted 2011-02-16; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: ACNE VULGARIS
MeSH Terms: conditions — Acne Vulgaris | interventions — Doxycycline; Equol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral antibiotic plus soy extract (Active Comparator)
  Interventions: Drug: Doxycycline and S-equol
- Oral antibiotic (Active Comparator)
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline and S-equol — Oral doxycycline and s-equol twice a day
  Arms: Oral antibiotic plus soy extract
Drug: Doxycycline — ORAL DOXYCYCLINE TWICE A DAY
  Arms: Oral antibiotic

SUMMARY:
The purpose of this study is to evaluate a novel, combination product for the treatment of acne vulgaris in females

ELIGIBILITY:
Inclusion Criteria:

* Healthy females 13 years of age or older
* Non-pregnant, non-lactating females
* Signed written informed consent form
* Must be able to understand and be willing to follow all study instructions
* Have a clinical diagnosis of acne vulgaris

Exclusion Criteria:

* Female subjects who are pregnant or nursing
* Any concomitant dermatologic condition that may affect outcome measures
* Concurrent use of any other medication to treat acne vulgaris
* Have a history or clinical evidence of any other active acute or chronic medical disease or condition considered by the principal investigator as unsuitable for the study
* Are currently using any other investigational agent or device
* Have participated in any other clinical study within 90 days prior to enrollment
* Employees or family members of sponsor or research site

Ages: 13 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
The mean number of Inflammatory Lesions on the face at the beginning and end of treatment | 12 weeks
  The number of inflammatory lesions will be counted by a trained investigator at the beginning and end of treatment.

SECONDARY OUTCOMES:
The mean number of Comedones will be evaluated at the beginning and end of treatment | 12 weeks
  A trained investigator will count the number of comedones at the beginning and end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Berlin, MD, Principal Investigator — Study Protocol, Inc.
Locations (2):
- United States (2):
  - Palos Verdes Dermatology Associates, Rolling Hills Estates, California
  - Berlin Center, Boynton Beach, Florida